CLINICAL TRIAL: NCT02324140
Title: The Impact of Genetic Variability on Perioperative Morbidity and Mortality. Substudy: Inflammatory Response in Patients Undergoing Aortic Valve Replacement.
Brief Title: Inflammatory Response in Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09_2
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Inflammation; Systemic Inflammatory Response Syndrome; Thoracic Surgery; Aortic Valve Stenosis
MeSH Terms: conditions — Inflammation; Systemic Inflammatory Response Syndrome; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Minimized extracorporeal circulation: Patients with severe aortic valve stenosis undergoing surgical aortic valve replacement using the minimized extracorporeal circulation (MECC, group 1)
  Interventions: Other: Whole blood analysis
- Conventional extracorporeal circulation: Patients with severe aortic valve stenosis undergoing surgical aortic valve replacement using the conventional extracorporeal circulation (CECC, group 2)
  Interventions: Other: Whole blood analysis
- Transcatheter aortic valve implantation, transfemoral access: Patients with severe aortic valve stenosis undergoing transcatheter aortic valve implantation using the transfemoral access route
  Interventions: Other: Whole blood analysis
- Transcatheter aortic valve implantation, transapical access: Patients with severe aortic valve stenosis undergoing transcatheter aortic valve implantation using the transapical access route
  Interventions: Other: Whole blood analysis

INTERVENTIONS:
Other: Whole blood analysis — In all fours groups of patients we investigate inflammatory and antiinflammatory response to the surgical and interventional treatment by analyzing changes in the concentration of interleukins, C-reactive protein, soluble CD62L and HLA-DR.

SUMMARY:
The study investigates inflammatory and antiinflammatory response in patients with severe aortic valve stenosis needing either surgical treatment (surgical aortic valve replacement) or interventional cardiology treatment (transcatheter aortic valve implantation using the transfemoral access route or the transapical access route).

DETAILED DESCRIPTION:
Background

Surgical and interventional therapy for aortic valve stenosis exposes the patients to a immune reaction, which is different depending on the type of the treatment. In this study, the investigators would like to better understand the inflammatory and antiinflammatory response in this patient population by monitoring the perioperative cytokine response (interleukins), the human leukocyte antigen expression (HLA-DR) and assessing soluble plasma factors (CD62L) involved in inflammatory processes.

Objective

Characterisation of inflammatory and antiinflammatory response in patients receiving aortic valve prosthesis selected for different treatment options.

Methods

Whole blood analysis at different time points (preoperatively, 4 / 24 /48 hours postoperatively) for different inflammatory and antiinflammatory markers: IL-6, IL-8, IL-10, CRP, TNF, soluble CD62L.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Severe aortic valve stenosis
* Surgical aortic valve replacement
* Transcatheter aortic valve implantation
* No previous inflammatory condition

Exclusion Criteria

* Missing informed consent
* Treatment with corticosteroids
* Treatment with antibiotics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic valve stenosis selected for surgical aortic valve replacement or transcatheter aortic valve implantation.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Inflammatory response, as determined by whole blood analysis of inflammatory biomarkers (IL-6, CRP, TNF alpha, CD62L) | Perioperative period ending after 48 hours postoperatively

SECONDARY OUTCOMES:
Anti-inflammatory response, as determined by whole blood analysis of inflammatory biomarkers (IL-8, IL-10) | Perioperative period ending after 48 hours postoperatively
In-hospital mortality | In-hospital treatment until discharge (7-10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Stüber, MD, Prof., Study Director — Dep. Anesthesiology and pain Therapy
Locations (1):
- Dep. Anesthesiology and Pain Therapy, Bern, Switzerland